CLINICAL TRIAL: NCT00529230
Title: Prevalence of Secondary Hypogonadism in Male Patients on Chronic Opioid Therapy for Cancer-Related Pain Syndromes
Status: Terminated | Type: Observational
Why Stopped: Low accrual rate.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: ID01-451
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Advanced Cancer; Hypogonadism; Pain
Keywords: Advanced Cancer; Chronic Opioid Therapy; Secondary Hypogonadism; Cancer-Related Pain Syndromes; Questionnaire
MeSH Terms: conditions — Hypogonadism; Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood draws to assess gonadal function.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic opioid therapy + Gonadal function: Males on chronic opioid therapy for cancer-related pain syndromes
  Interventions: Behavioral: Questionnaire; Other: Blood draws to assess gonadal function

INTERVENTIONS:
Behavioral: Questionnaire — A set of questionnaires regarding sexual function, physical and psychological symptoms.
Other: Blood draws to assess gonadal function — Testosterone, FSH, and LH levels at study onset.

SUMMARY:
Primary Objective:

1. To determine the prevalence of secondary hypogonadism in male patients on chronic opioid therapy for cancer-related pain syndromes.

Secondary Objective:

1. To determine the degree of sexual dysfunction, fatigue, and depression prevalent in male patients on chronic opioid therapy for cancer-related pain syndromes.

DETAILED DESCRIPTION:
Studies have shown that non-cancer patients taking opioid pain medication for a long period of time can have decreased libido and decreased sexual function.

Individuals may be asked to take part in this study even if they have not taken opioid pain medications in the last twelve months. These individuals would also be enrolled to learn if long-term treatment of cancer-related pain with opioid medications results in decreased sex hormones, decreased sex drive, and increased fatigue or depression.

Participants in this study will be asked to complete a set of questions about their sexual functions, physical symptoms, and psychological symptoms such as fatigue and depression. It will take about 25 minutes to complete the questionnaires.

Participants will have blood drawn (about 2 teaspoons of blood) to test their sex hormone level. Participants who are identified as having low sex hormone level (hypogonadism) will be referred to an endocrinologist for standard hormone replacement therapy.

This is a one-time evaluation, no follow-up visit or questionnaires are required.

This is an investigational study. A total of 108 individuals will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic pain greater than one year.
2. Male.
3. Cancer status must be stable or in remission. For this study, "stable disease" is defined as identifiable disease at local or metastatic sites that has shown no progression over the previous 3 months and there has been no cancer treatment for ³ 3 months.
4. Patients must be on chronic opioid therapy on a continuous basis in the preceding twelve months with a Morphine Equivalent Daily Dose (MEDD) ³ 200.
5. Age >/= 18. The questionnaires used in this study have been validated only in the adult population. In addition, some of the questionnaires contain questions of a sensitive nature and are not appropriate in the pediatric population.
6. Patients must be able to understand and sign the consent form.

Exclusion Criteria:

1. Patient who refuses to participate in the study or determined incapable of completing the research.
2. Patients with pre-existing hypopituitarism. Causes include certain tumors (pituitary adenomas, hypothalamic tumors), inflammatory diseases (granulomatous diseases), vascular diseases (postpartum necrosis, carotid aneurysm), traumatic/destructive events (prior surgery, trauma, or radiation), developmental anomalies, infiltration.
3. Patients who tare taking any drugs that may affect the hypothalamic-pituitary-gonadal axis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males on chronic opioid therapy for cancer-related pain syndromes.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2001-12-11 (Actual); Primary Completion 2004-02-19 (Actual); Study Completion 2004-02-19 (Actual)

PRIMARY OUTCOMES:
Prevalence of secondary hypogonadism in male patients on chronic opioid therapy for cancer-related pain syndromes | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajagopal, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States